CLINICAL TRIAL: NCT01427335
Title: Does Intravenous Calcium Infusion Effectively Prevent OHSS : a Randomised Controlled Trial
Brief Title: Calcium for Prevention of Ovarian Hyperstimulation Syndrome
Acronym: OHSS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Waleed El-khayat, Doctor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 192011
Record Dates: First submitted 2011-08-31; First posted 2011-09-01 (Estimated); Last update posted 2014-07-09 (Estimated); Status verified 2014-07

CONDITIONS: Ovarian Hyperstimulation Syndrome
Keywords: OHSS; ICSI; calcium injection
MeSH Terms: conditions — Ovarian Hyperstimulation Syndrome | interventions — Calcium; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- saline (Placebo Comparator): 0.9% saline intravenous infusion
  Interventions: Drug: 0.9 % saline
- calcium (Experimental): Calcium intravenous infusion
  Interventions: Drug: calcium

INTERVENTIONS:
Drug: calcium — intravenous infusion of 10 % calcium gluconate 10 mL in 200 mL of physiologic saline on the day of ovum pickup, day 1,day 2, and day 3 after ovum pickup were administered in study group.
  Intravenous infusion was performed within 30 minutes
  Other Names: Calcium intravenous infsuion
  Arms: calcium
Drug: 0.9 % saline — 0.9 % saline intravenous infusion
  Arms: saline

SUMMARY:
There are many protocols for prevention of ovarian hyperstimulation syndrome, intravenous calcium is a novel protocol. But still there is lack of evidence of it is real effect in prevention of OHSS & the mechanism of its action is still questionable . In the study the investigators try to search for the evidence for its effect & the real mechanism for its action.

DETAILED DESCRIPTION:
The study population will be divided into 2groups each containing 100 infertile couples candidate for ICSI.

Group (A)active group: administration of 10% Intravenous calcium gluconate 10 ml in 200 mL of physiologic saline on the day of ovum pickup, day 1,day 2, and day 3 after ovum pickup. Intravenous infusion was performed within 30 minutes.

Group (B): placebo group: administration of 200 mL of 0.9% saline on the day of ovum pickup, day 1,day 2, and day 3 after ovum pickup. Intravenous infusion was performed within 30 minutes

ELIGIBILITY:
Inclusion Criteria:

* infertile women aged 20 to 38 years.
* BMI ranged from 18 to 40.
* serum FSH within normal limits( 1-12IU /l)
* presented with ovarian response suggestive of being at risk of developing OHSS because of the presence of at least 15 follicles of 10 mm or greater on the day of hCG administration.

Exclusion Criteria:

* endocrinopathies.
* a systemic disease.
* using any medication (e.g., insulin-sensitizing drugs and GnRH antagonists.
* patients need coasting for high risk of OHSS.
* patients need cycle cancellation.
* severe male infertility requiring testicular sperm extraction.

Ages: 20 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2011-10; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
OHSS rate | 2 years
  ovarain hyperstimulation syndrome

SECONDARY OUTCOMES:
clinical pregnancy rate | 2 years
  positive pregnancy test and positive fetal heart beat after 6 weeks gestaional age

CONTACTS AND LOCATIONS:
Overall Officials: Waleed M El-Khayat, M.D., Principal Investigator — Cairo University
Locations (1):
- Kasr elini hospital, Cairo, Cario, Egypt

REFERENCES:
- [Derived] El-Khayat W, Elsadek M. Calcium infusion for the prevention of ovarian hyperstimulation syndrome: a double-blind randomized controlled trial. Fertil Steril. 2015 Jan;103(1):101-5. doi: 10.1016/j.fertnstert.2014.09.046. PMID 25552412